CLINICAL TRIAL: NCT07019155
Title: Longitudinal Study of Individuals and Families With Aberrations in DDX41 or Similar Cancer Predisposition Variants
Brief Title: Study of Individuals and Families With Aberrations in DDX41 or Similar Cancer Predisposition Variants
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002394; 002394-C
Record Dates: First submitted 2025-06-12; First posted 2025-06-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12-10

CONDITIONS: Germline Mutation; Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: DEAD-box helicase 41 (DDX41); germline mutations; MDS; AML; Germline Predisposition Syndromes; Hereditary Hematopoietic Malignancy; Cancer Predisposition
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Participants with confirmed aberrations that affect the DDX41 gene, DDX41 RNA, or DDX41 protein and who have a history of MDS/MPN/AML diagnosis
- Cohort 2: Participants with confirmed aberrations that affect the DDX41 gene, DDX41 RNA, or DDX41 protein and who do NOT have history of MDS/MPN/AML
- Cohort 3: Participants with confirmed aberrations in another HHM variant
- Cohort 4: Participants with confirmed absence of known HHM variants, and who have first or second degree relative with confirmed or suspected HHM variant(s) (control group)

SUMMARY:
Background:

Hereditary hematopoietic malignancy (HHM) syndromes are a group of inherited disorders that raises the risk of blood cancers. Many people with HHMs have changes in a gene (DDX41) that makes it more likely that they will develop myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), or other cancers. This natural history study will explore the link between HHM syndromes and these diseases.

Objective:

To study the link between HHM and MDS/AML.

Eligibility:

People aged 1 month and older with HHM. Relatives with HHM are also needed.

Design:

Participants aged 3 years and older will have 1 initial clinic visit with the option to follow-up annually. They will undergo these procedures:

They will have a physical exam with blood and urine tests.

They may give samples of saliva, stool, nails, and skin.

Their ability to do normal activities will be reviewed.

Some may have a bone marrow biopsy: A tissue sample will be drawn from inside a bone.

They may answer questions about their health and family medical history.

Participants younger than 3 years, and those who cannot come to the clinic, will be contacted by phone or email. Their samples may be collected locally and sent to researchers.

For participants who have changes in their DDX41 gene: Researchers will contact them or their primary care provider once a year for 10 years. Researchers will check on participants health and collect any new test results. Some may be asked to send new samples.

Participants who do not have changes in their DDX41 gene may be contacted yearly, or less often, for 10 years.

Some participants may be asked to return to the clinic if needed.

DETAILED DESCRIPTION:
Background:

* Growing awareness of germline predisposition syndromes raises questions about how to best identify, test, and manage individuals carrying germline variants with 1.5%-6.1% of individuals with hematologic malignancies carrying an identified aberration.
* Germline mutations in DEAD-box helicase 41 (DDX41) were first identified as a susceptibility to myeloid neoplasms in 2015 and have been described in up to 6.1% in myelodysplastic syndromes (MDS)/acute myeloid leukemia (AML) patients.
* Germline DDX41 variants are associated with a distinct subtype of myeloid neoplasms, marked by familial predisposition, male predominance, and several commonly commutated somatic genes such as AXL1, EZH2, SRSF2, CUX1 and TP53, and a few underrepresented mutations such as TET2, SF3B1 and NPM1.
* Somatic deleterious variants of the second allele in patients with DDX41 germline variants leads to the onset of multiple lineage cytopenias at a mean age of 66 years (range 50-85 years), followed by the development of a hematologic malignancy.
* The myeloid malignancy associated with DDX41 variants is generally responsive to standard upfront chemotherapy. However, relapses are common and the median survival for individuals with MDS/AML secondary to germline DDX41 variants is consistent with de novo AML at approximately 5.2 years.
* In cases of familial MDS/AML associated with DDX41, the family history may appear negative due to failure to recognize the disorder in family members, reduced penetrance, or late onset of disease.
* Other germline variants in genes such as, but not limited to, CEBPA, CHEK2, ETV6, Fanconi genes, GATA2, RUNX1, and short telomere syndrome associated genes also confer hereditary hematopoietic malignancy (HHM) risk and may induce downstream effects on DDX41. Combinations of variants may exhibit variable clinical presentations, phenotypic associations, therapy responses, and treatment outcomes.
* Currently there are no biomarkers or assays to predict which patients with known HHM variants will progress to a malignancy, and many patients present with a myeloid malignancy as their initial manifestation of a germline syndrome.

Objective:

-To estimate the event free survival (EFS) in individuals with DEAD-box helicase 41 (DDX41) aberrations

Eligibility:

* Age > 1 month old
* Must have confirmed aberrations that affect the DDX41 gene, DDX41 RNA, or DDX41 protein or confirmed aberrations in another HHM variant

or

must have confirmed absence of HHM variants and have first or second degree relative with confirmed or suspected HHM variant(s)

-Must have an identified medical provider outside NIH who manages care, and any diagnostic findings provided by this study.

Design:

* This is a natural history and biospecimen analysis protocol for participants with aberrations in DDX41 or other HHMs and relatives of individuals with aberrations in DDX41 or other HHMs.
* We will perform comprehensive research analysis to understand the biology of HHM variants that contributes to dysregulation in hematopoietic differentiation and maturation blocks leading to dysplasia, cytopenia, and disease progression, so that these may be exploited for novel therapeutic targeting strategies.
* Diagnostic testing will be performed as is routine for these participants in addition to planned research correlative analyses. Follow-up will occur approximately annually to assess status and survival.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age > 1 month old.
* Participants with history of aberrations that affect the DDX41 gene, DDX41 RNA, or DDX41 protein (Cohorts 1-2)

OR

Participants with history of aberrations in another HHM variant (Cohort 3)

OR

Participants with history of absence of HHM variants, who have first or second degree relative with history of confirmed or suspected HHM variant(s) per participant report (Cohort 4).

* Participants must have an identified healthcare provider outside of NIH who manages participant care, and any diagnostic clinical findings provided by this study.
* Ability of participant or parent/guardian to understand and the willingness to sign a written consent document.

EXCLUSION CRITERIA:

None.

Ages: 1 Month to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with aberrations in DDX41 or other HHMs and relatives of individuals with aberrations in DDX41 or other HHMs.
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2035-06-15 (Estimated); Study Completion 2035-06-15 (Estimated)

PRIMARY OUTCOMES:
To estimate the EFS in individuals with DEAD-box helicase 41 (DDX41) aberrations | Up to 10 years
  Describe the EFS separately for Cohort 1 and Cohort 2. Kaplan-Meier plots will be generated, five and 10-year EFS will be reported, along with 95% confidence intervals for each Cohort separately.

SECONDARY OUTCOMES:
To define the OS in individuals with DDX41 aberrations | Up to 10 years
  Describe the overall survival of participants for Cohorts 1 and 2 separately utilizing Kaplan-Meier plots. Five and 10-year OS will be reported, along with 95% confidence intervals.
To identify secondary commonly co-mutated somatic or germline variants as well as underrepresented mutations that may impact clinical presentation, disease severity, progression to malignancies. | Up to 10 years
  Co-mutations will be descriptively tabulated. The proportion of participants with each co-mutation will be described for Cohorts 1, 2, 3, and 4 separately, along with 95% confidence intervals per the exact Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Yun Pai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002394-C.html